CLINICAL TRIAL: NCT02774915
Title: Outcome of Pregnancy Associated Breast Cancer (PABC) in Saudi Arabia ; Prospective Cohort Study.
Brief Title: Outcome of Pregnancy and Breast Cancer
Acronym: Pregnancy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Guard Health Affairs (Other Government)
Responsible Party: Sponsor
Other Study IDs: RC12/153/R
Record Dates: First submitted 2016-03-31; First posted 2016-05-17 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2016-05

CONDITIONS: Pregnancy; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Investigators are interested to explore the clinical and pathological characteristics of breast cancer with pregnancy, maternal age at the time of diagnosis of breast cancer during pregnancy, median gestational age at diagnosis, the level of the tumor differentiation patients present with, during pregnancy, and the hormonal-receptor status. Investigators plan to collect prospective quality research databases that could provide further important information concerning this condition and serve in both short- and long-term sequelae in mother and fetus.

DETAILED DESCRIPTION:
Breast cancer is classified as pregnancy-associated if it is diagnosed during pregnancy or within one year of delivery . About 3% of all breast cancers are diagnosed during pregnancy . The average age at diagnosis for patients with PABC is 32-38 years .A painless mass is palpated by the patient in 90% of reported cases .The incidence of breast cancer is the same in pregnant women as nonpregnant women in the general population.

Breast cancer is the most common malignancy affecting women world wide. More than one million cases diagnosed annually. One in ten of all new cancers diagnosed worldwide each year is a cancer of the female breast, and it is the most common cancer in women in both developing and developed areas. It is also the principal cause of death from cancer among women globally. Similar applied to Saudi Arabia. More over, cancer registry suggested an increase in incidence over the years with median age of 67 years old. The same applied for other Arab regions. Recently, women in Arab regions postpone their first pregnancy which may increase the risk for pregnancy associated breast cancer.

The physiologic changes that take place in the breast during pregnancy can contribute to a delay in the diagnosis of PABC. In preparation for lactation, a women's breast size will nearly double in size and weight. The influence of estrogen and progesterone cause an increase in blood flow and fat, resulting in an increase in the size of milk-producing glands. Some women may begin to leak colostrum by 25 weeks gestation. Irritation of the breast ducts caused by rapid tissue growth may cause a bloody discharge, which usually is a benign condition. The areola also may increase in size and become darker in color. In addition, Montgomery tubercles, small nodules surrounding the areola, will produce a fluid to lubricate and cleanse the nipple in preparation for nursing.

Breast cancer associated with pregnancy presents to the clinician with particular challenges at diagnosis and management level. The diagnosis may be delayed and difficult owing to the physiological changes within the breast and limitations on investigations. Moreover once a diagnosis has been confirmed and staging completed, options for treatment will be influenced by the need to give optimal treatment to the mother whilst minimizing risks to the fetus. The particular challenges faced both in the initial diagnosis and management of women with pregnancy-associated breast cancer will be assessed in this study.

Recent studies suggest that, when matched for age and stage, the prognosis of pregnancy-associated breast cancer is comparable to non-pregnancy-associated breast cancer. However, the risk for breast cancer recurrence associated with subsequent pregnancies in this population is not clear. Although there is data showing no increase in the risk of recurrence for women who become pregnant after breast cancer treatment, pregnancy-associated breast cancer may be a distinct clinical category where subsequent pregnancies after treatment may confer an increased risk of recurrent disease9.

There is a lack of controlled data concerning the management of pregnancy-associated breast cancer, both locally and globally.

Investigators plan in this study to assess and document the clinical presentation, diagnosis, treatment, prognostic factors, and routine clinical management of pregnant ladies diagnosed with breast cancer in Saudi Arabia. Data base through data collection on all information related to breast cancer patients with pregnancy will be performed across detailed interview and chart review at all specialized clinic in the National Guard. All patients seen within the coming 5 years will be enrolled in this study.

Investigators are interested to explore the clinical and pathological characteristics of breast cancer with pregnancy, maternal age at the time of diagnosis of breast cancer during pregnancy, median gestational age at diagnosis, the level of the tumor differentiation patients present with, during pregnancy, and the hormonal-receptor status. Investigators plan to collect prospective quality research databases that could provide further important information concerning this condition and serve in both short- and long-term sequelae in mother and fetus.

ELIGIBILITY:
Inclusion Criteria:

• All pregnants with breast cancer will be included in this study

Exclusion Criteria:

• Refusal of pregnant women with 2nd or 3rd trimester to receive chemotherapy, will be excluded

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study design approach is a cohort study, which planned to recruit all patients attend the breast cancer clinic, interview in details, assessed and followed prospectively for 5 years from the time of diagnoses or till death occurs, whichever occurred first.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2014-11; Primary Completion 2019-11 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
To explore the characteristics of pregnancy associated breast cancer (PABC), maternal and fetal outcome of the pregnancy. | 5 years
Prevelance and outcome | 5 years
  • To determine the prevalence and incidence of breast cancer in pregnancy
prevalence and outcome | 5 years
  • To measure the prognostic outcomes of at mother and fetus level in breast cancer with pregnancy
prevalence and outcome | 5 years
  • To describe the pathological characteristics of breast cancer when it concomitantly present with pregnancy
prevalence and outcome | 5 years
  • To assess the sensitivity and specification of diagnostic procedure.

SECONDARY OUTCOMES:
Long outcome | 5 years
  * To measure the outcome of newborn after 1st and 5th year.
Long outcome | 5 years
  • To assess the outcome of breast cancer after 5 years from diagnosis

CONTACTS AND LOCATIONS:
Locations (1):
- King Abdul Aziz Medical City for National Guard Health Affairs, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No